CLINICAL TRIAL: NCT07300176
Title: Observation of the Effects of Virtual Reality-Assisted Intraoperative Sensory Modulation on Postpartum Depression, Cognitive Function, and the Kynurenine Pathway
Brief Title: Virtual Reality-Assisted Intraoperative Sensory Modulation on Postpartum Depression and the Kynurenine Pathway
Acronym: VR effect
Status: Active, not recruiting | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: tufantez2025
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Virtual Reality; Postpartum Depression (PPD); Kynurenine Pathway and Its Metabolites; Pregnancy; Satisfaction
Keywords: Postpartum Depression; Kynurenine Pathway; Cesarean Section; Sensory Modulation; Virtual Reality
MeSH Terms: conditions — Depression, Postpartum; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (VR group, n = 49):: Patients who underwent cesarean section under spinal anesthesia and received intraoperative virtual reality (VR) intervention via a VR headset to provide sensory modulation.
- Group 2 (Control group, n = 49): Patients who underwent cesarean section under spinal anesthesia and received standard clinical care without any VR application

SUMMARY:
The research will be conducted as a prospective, observational, and comparative study with 98 pregnant volunteers aged 18-45 at Düzce University Faculty of Medicine. Participants will be divided into a VR group and a control group. Data will be collected using STAI-I, EPDS, NRS scales, and biochemical analyses (tryptophan, kynurenine, etc.).

Upon completion, the project is expected to contribute to non-pharmacological approaches and new care protocols for reducing postpartum depression.

DETAILED DESCRIPTION:
1. Ethics Approval, Study Design and Sample Size This study was conducted after obtaining approval from the Düzce University Non-Interventional Clinical Research Ethics Committee (Date: 10.11.2025, Decision No: 2025/285) and with the support of the Düzce University Scientific Research Projects (BAP) Coordination Unit (Project No: [Project Number]). The study was carried out in accordance with the principles of the Declaration of Helsinki.

   The research was planned as a prospective, observational study. It was conducted between October 2025 and August 2026 at Düzce University Health Application and Research Center in patients undergoing elective cesarean section.

   The sample size was calculated using the G*Power software (Version 3.1.9.4), based on an ANOVA for repeated measures with between-subjects factors. Assuming 80% power (1-β), a Type I error rate of 5% (α = 0.05) and a medium effect size (f = 0.25), the minimum required total sample size was calculated as 98 for two groups and two repeated measurements (postpartum week 1 and week 6 depression scores), corresponding to 49 participants per group.

   Written informed consent was obtained from all participants after they were given detailed information about the aim and procedures of the study.

   ________________________________________
2. Study Population and Eligibility Criteria Inclusion criteria

   * Pregnant women scheduled for elective cesarean section
   * Age between 18 and 45 years
   * ASA physical status I-II
   * No contraindication to spinal anesthesia
   * Signed written informed consent Exclusion criteria
   * Anticipated need for postoperative intensive care unit (ICU) admission
   * History of psychiatric or neurological disease
   * Visual or auditory impairment
   * Severe preeclampsia, eclampsia, or HELLP syndrome
   * Perinatal loss (postpartum neonatal death)
   * History of convulsions or epilepsy
3. Study Procedure and Grouping

A total of 98 patients who met the eligibility criteria were included and, in line with the observational design, were allocated into two groups:

* Group 1 (VR group, n = 49): Patients who underwent cesarean section under spinal anesthesia and received intraoperative virtual reality (VR) intervention via a VR headset to provide sensory modulation.
* Group 2 (Control group, n = 49): Patients who underwent cesarean section under spinal anesthesia and received standard clinical care without any VR application.

All patients underwent routine preoperative anesthetic evaluation in the anesthesia outpatient clinic. On the day of surgery, the State-Trait Anxiety Inventory-State form (STAI-I) was administered intraoperatively to assess anxiety levels.

In the operating room, after spinal anesthesia was performed and the sterile field was established, patients in Group 1 were fitted with a VR headset displaying preselected, nature-based, relaxation-oriented virtual reality content. The VR application was maintained continuously throughout the procedure until completion of skin closure, except for the moment of first maternal-infant contact. Patients in Group 2 received only standard clinical care and no VR headset was applied.

* Data Collection Tools and Measurements Study data were collected using demographic information forms, validated psychometric scales, and biochemical analyses.

  4.1. Anxiety Assessment Patients' state anxiety levels were assessed using the State-Trait Anxiety Inventory-State form (STAI-I), originally developed by Spielberger et al. (1970) and adapted and validated in Turkish by Öner and Le Compte (1983). This self-report instrument consists of 20 items that evaluate the individual's current emotional state and intensity of anxiety at the time of assessment.

  4.2. Postpartum Depression Assessment Postpartum depression was screened using the 10-item Edinburgh Postnatal Depression Scale (EPDS), developed by Cox et al. (1987) and validated in Turkish by Engindeniz et al. (1996). The EPDS was administered at postpartum week 1 and week 6 to evaluate depressive symptoms.

  4.3. Patient Satisfaction Assessment Patient satisfaction with the operative experience was evaluated at the end of surgery using a Numerical Rating Scale (NRS). The NRS is a commonly used instrument providing a numerical rating from 0 (not satisfied at all) to 10 (completely satisfied).

  4.4. Biochemical Measurements For biochemical analyses, residual plasma samples obtained from routine preoperative and 24-hour postpartum blood tests were used. After collection, blood samples were centrifuged under appropriate conditions, and plasma aliquots were stored at -80°C until analysis. Plasma levels of kynurenine, kynurenic acid, tryptophan and quinolinic acid were measured using commercially available enzyme-linked immunosorbent assay (ELISA) kits, according to the manufacturer's instructions.

  ________________________________________
* Statistical Analysis Statistical analyses were performed using IBM SPSS Statistics (Version XX, IBM Corp., Armonk, NY, USA). The normality of continuous variables was assessed using the Kolmogorov-Smirnov or Shapiro-Wilk tests, as appropriate. For between-group comparisons, the independent samples t-test was used for normally distributed continuous variables, and the Mann-Whitney U test for non-normally distributed variables. Categorical variables were compared using the chi-square test or Fisher's exact test when expected cell counts were small.

Within-group changes over time (preoperative vs. postpartum measurements) were analyzed using the paired samples t-test for normally distributed data or the Wilcoxon signed-rank test for non-normally distributed data. A two-sided p value < 0.05 was considered statistically significant for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women scheduled for elective cesarean section
* Age between 18 and 45 years
* ASA physical status I-II
* No contraindication to spinal anesthesia
* Accepted for VR equipment usage during operation.
* Signed written informed consent

Exclusion Criteria:

* Anticipated need for postoperative intensive care unit (ICU) admission
* History of psychiatric or neurological disease
* Visual or auditory impairment
* Severe preeclampsia, eclampsia, or HELLP syndrome
* Perinatal loss (postpartum neonatal death)
* History of convulsions or epilepsy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of pregnant women scheduled for elective cesarean section under spinal anesthesia. Participants will be recruited from the obstetrics and gynecology department of the participating hospital. Eligible individuals must be between 18 and 45 years of age, carrying a singleton pregnancy, clinically stable for regional anesthesia and accepted for VR equipment usage during operation.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Edinburgh Postnatal Depression Scale (EPDS) | up to 6 weeks
  The Edinburgh Postnatal Depression Scale (EPDS) will assess depressive symptoms related to the peripartum period. Measurements will be obtained preoperatively and after the intraoperative VR application. Changes in EPDS scores (numbers 0-30 ) will help determine whether VR reduces depressive affect during the surgical experience.
Change in State-Trait Anxiety Inventory-State (STAI-I) score | up to 6 weeks
  The State-Trait Anxiety Inventory-State (STAI-I) score ( number 16-80) will be used to assess changes in acute anxiety levels in pregnant patients undergoing cesarean section under spinal anesthesia. Scores will be recorded immediately before the intraoperative VR intervention and again during the procedure. A reduction in STAI-I score following VR exposure will indicate decreased anxiety.

SECONDARY OUTCOMES:
Biochemical Levels of Kynurenine Pathway Metabolites | up to 6 weeks
  Blood samples will be collected before the surgical procedure and postoperatively to quantify serum levels of key metabolites in kynurenine (ng/mL), kynurenic acid (ng/mL), tryptophan (ng/mL), and quinolinic acid (ng/mL) . Analytical methods (e.g., HPLC or LC-MS/MS) will be used to measure changes induced by the VR intervention. These biomarkers will help evaluate the physiological stress response and potential neuromodulatory effects of VR.
Patient Satisfaction Numerical Rating Scale score | up to 6 weeks
  Patient satisfaction will be assessed postoperatively using the Numerical Rating Scale (Number 0-10), where higher scores indicate greater satisfaction with the anesthesia and intraoperative experience. This secondary outcome evaluates whether VR improves overall comfort and satisfaction during spinal anesthesia for cesarean delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: 10/12/2025 (start date) 10/12/2030 (end date)
Access Criteria: All the people